CLINICAL TRIAL: NCT00094445
Title: Phase II Trial of Curcumin in Patients With Advanced Pancreatic Cancer
Brief Title: Trial of Curcumin in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sabinsa Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0009; 1R21CA104337 (NIH); NCI-2012-01309 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2004-10-18; First posted 2004-10-19 (Estimated); Results first posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Pancreatic Neoplasms; Adenocarcinoma
Keywords: Pancreatic Cancer; Adenocarcinoma of the pancreas; Alternative therapy; Pancreas; Pancreatic Neoplasm; Cancer of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma | interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Curcumin (Experimental): Oral curcumin daily for eight weeks, starting dose 8 gm per day.
  Interventions: Drug: Curcumin

INTERVENTIONS:
Drug: Curcumin — Starting dose 8 gm orally per day for 8 weeks. If patient experiences grade III toxicity, dose held and restarted with a 50% dose reduction after resolution of toxicity to </= Grade I. Patients with grade IV toxicity will discontinue treatments. Patients with </= grade I toxicity may have a 25% dose increase at each four-week period. Patients will continue on treatment until disease progresses, unless Grade III toxicity supervenes.
  Other Names: diferuloyl methane

SUMMARY:
The goal of this clinical research study is to learn if treatment with curcumin can help shrink or slow the growth of pancreatic cancers. The effect of curcumin on the way pancreatic cancer cells function and the safety of treatment with curcumin will also be studied.

DETAILED DESCRIPTION:
Curcumin, a yellow substance extracted from the plant Curcuma longa, is commonly used as a food additive. It is a natural anti-inflammatory compound and has shown anti-tumor activity in the laboratory. During this study, you will receive much higher doses of curcumin than can be obtained from the diet.

During the study, you will receive curcumin by mouth every day. You will be required to take up to 16 pills per day each morning. Every 8-week period you take curcumin is considered a "course" of treatment. The number of courses you receive depends on how you are responding to treatment. You can continue treatment as long as the disease does not get worse. If the disease gets worse or you experience any intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

You will be given a questionnaire to complete at the beginning of the study and once a week while you are on therapy to help the medical staff understand how the different symptoms from your disease are affecting you. This questionnaire, which should take about 5 minutes to complete, can be done over the telephone or with the help of one of the study staff during your visits.

At the end of each course of treatment (every 8 weeks), you will have a physical exam and the tumor will be re-evaluated using CT scans and/or blood (about 2 tablespoons) tests.

This is an investigational study. Curcumin is a commercially available substance, which is commonly used as a food additive. Up to 50 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has pathologically confirmed adenocarcinoma of the pancreas that is not amenable to curative surgical resection (includes locally advanced, metastatic, or recurrent disease). Histology must be confirmed by the pathology department of the investigational center.
2. The patient has a Karnofsky Performance Status of greater than or equal to 60 at study entry.
3. The patient has given informed consent.
4. The patient is at least 18 years of age.
5. The patient has adequate hematologic function as defined by an absolute neutrophil count greater than or equal to 1,500/mm3, platelet count greater than or equal to 100,000/mm3.
6. The patient has adequate hepatic function as defined by a total bilirubin less than or equal to 2.0 X ULN, alkaline phosphatase, AST and/or ALT less than or equal to 5 X ULN, and creatinine less than or equal to 2.0 mg/dL.
7. The patient has measurable disease.
8. The patient agrees to use effective contraception if procreative potential exists.

Exclusion Criteria:

1. The patient has a history of treated or active brain metastases, carcinomatous meningitis, an uncontrolled seizure disorder, or active neurological disease.
2. The patient has received prior radiation. Patients with measurable disease outside the radiation port or documented disease progression of previously irradiated measurable disease are eligible. Patient must be greater than or equal to four weeks post-therapy and have recovered from all toxicities.
3. The patient has an unstable medical condition according to the investigator, including uncontrolled diabetes mellitus or hypertension; active infections requiring systemic antibiotics, antivirals, or antifungals, unstable CHF, uncontrolled arrythmias, or unstable coagulation disorders.
4. The patient is pregnant (confirmed by serum Beta-HCG) or is breast feeding.
5. The patient has received an investigational agent(s) within four weeks of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Subbiah, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Background] Aggarwal BB, Kumar A, Bharti AC. Anticancer potential of curcumin: preclinical and clinical studies. Anticancer Res. 2003 Jan-Feb;23(1A):363-98. PMID 12680238
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: November 12, 2004 to November 11, 2010. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: 1 participant did not receive treatment due to screen failure, patient withdrew the consent
Period: Overall Study
Arm/Group | Curcumin
Started | 50
Completed | 44
Not Completed | 6
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1
Not completed — Progressive Disease | 2

BASELINE CHARACTERISTICS:
Arm/Group | Curcumin
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 65 [40 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Six-Month Participant Survival
Description: Number of participants followed from baseline (date of randomization) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months.
Time Frame: Baseline to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Curcumin
Number analyzed (Participants) | 44
Participants | 7

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Curcumin
Serious Adverse Events (participants affected / at risk) | 9/44
Other Adverse Events (participants affected / at risk) | 6/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Curcumin (N=44)
GI hemmorhage (Gastrointestinal disorders) | 1
Chest pain (Cardiac disorders) | 1
Multiple pulmonary emboli (Cardiac disorders) | 1
chronic cancer progression (Gastrointestinal disorders) | 1
abdomen pain (Gastrointestinal disorders) | 2
acute renal failure (Renal and urinary disorders) | 1
metastasis (Gastrointestinal disorders) | 1
weakness (General disorders) | 1
dehydration (General disorders) | 1
slurred speech (Nervous system disorders) | 1
confusion (Nervous system disorders) | 1
anorexia (Metabolism and nutrition disorders) | 3
non-neutropenic fever (General disorders) | 1
musculoskeletal (Musculoskeletal and connective tissue disorders) | 1
ascites (Gastrointestinal disorders) | 1
constipation (Gastrointestinal disorders) | 1
mood alteration (Nervous system disorders) | 1
vomiting (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Chronic colocutaneous fistula (Gastrointestinal disorders) | 1
abdominal wall abscess (Gastrointestinal disorders) | 1
infection (Infections and infestations) | 1
atrial fibrillation (Cardiac disorders) | 1
atrial flutter (Cardiac disorders) | 1
indigestion (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Curcumin (N=44)
edema (Skin and subcutaneous tissue disorders) | 4
vomiting (Gastrointestinal disorders) | 2
nausea (Gastrointestinal disorders) | 2
abdomen (Gastrointestinal disorders) | 1
depression (Nervous system disorders) | 1
Fatigue (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No